CLINICAL TRIAL: NCT05113615
Title: Daily Dosing of Tiotropium and Tolerance to Bronchoprotection Against Methacholine Challenge
Brief Title: Regular Use Tiotropium and Tolerance to Bronchoprotection in Mild Asthma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Don Cockcroft, Professor, University of Saskatchewan
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Bio ID 2985
Record Dates: First submitted 2021-10-28; First posted 2021-11-09 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Asthma
Keywords: tiotropium; bronchoprotection; tolerance; methacholine PD20
MeSH Terms: conditions — Asthma | interventions — Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tiotropium bromide (Active Comparator): tiotropium bromide inhaler (Spiriva Respimat) will be used once daily (2 puffs) for a total of 8 days
  Interventions: Drug: Tiotropium Bromide
- Matching placebo (Placebo Comparator): matching placebo inhaler will be used once daily (2 puffs) for a total of 8 days
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: Tiotropium Bromide — respimat inhaler 2.5mcg/puff
  Other Names: Spiriva Respimat
  Arms: tiotropium bromide
Drug: Matching placebo — matching placebo Respimat inhaler
  Arms: Matching placebo

SUMMARY:
The study will assess if regular use of tiotropium (i.e. daily) results in loss of bronchoprotection against methacholine induced bronchoconstriction in those with mild asthma.

DETAILED DESCRIPTION:
A single dose of an inhaled muscarinic antagonist will protect against methacholine induced bronchoconstriction and increase the dose of methacholine required to cause bronchoconstriction about 4 doubling doses. Beta agonist bronchodilators also shift the dose response curve to the right but the protection against methacholine induced bronchoconstriction is lost (i.e. tolerance develops) with regular use. This study will determine if bronchoprotection is lost following regular use of tiotropium.

This will be a randomized, double-blind placebo controlled study to assess the development of tolerance following regular use of tiotroium in a population of mild asthmatics.

Tiotropium will be administered at the clinically recommended dose (5mcg/day) for a total of 8 days. Methacholine challenges will be performed at baseline (pre-treatment), at one hour post first dose and on day 8, one hour after the final dose. The same will dosing schedule and assessments will occur with an identical placebo inhaler.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of asthma
* asthma is currently well controlled using only occasional bronchodilators
* baseline lung function (FEV1) is greater than 65% of the predicted value
* exhibit bronchoconstriction to inhaled methacholine at a dose of 200mcg or less

Exclusion Criteria:

* women who are pregnant or breastfeeding.
* diagnosis of another lung condition or medical condition that would pose a risk to the participant if enrolled in the study
* current smokers of nicotine products (e.g., cigarettes).
* users of cannabis or other inhaled recreational products (e.g., e-cigarettes or other vaping products) on a daily basis
* respiratory infection within 4 weeks of entering the study
* use of any anticholinergic agent within 30 days prior to the beginning of the study (e.g., ipratropium or the study treatment tiotropium).
* known hypersensitivity to tiotropium bromide or components of tiotropium formulation (e.g., benzalkonium chloride), to atropine or its derivatives.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2022-05-06 (Actual); Study Completion 2022-05-06 (Actual)

PRIMARY OUTCOMES:
Methacholine PD20 | pre treatment
  dose of methacholine required to induce a 20% fall in FEV1 (volume of air forcefully exhaled in the first second following a full inhalation)
Methacholine PD20 | one hour post first dose
  dose of methacholine required to induce a 20% fall in FEV1 (volume of air forcefully exhaled in the first second following a full inhalation)
Methacholine PD20 | one hours post final dose
  dose of methacholine required to induce a 20% fall in FEV1 (volume of air forcefully exhaled in the first second following a full inhalation)

CONTACTS AND LOCATIONS:
Overall Officials: Don Cockcroft, MD, Principal Investigator — University of Saskatchewan
Locations (1):
- Asthma Research Lab University of Saskatchewan Room 346 Ellis Hall, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No